CLINICAL TRIAL: NCT04474275
Title: The Effect of the Mode of Delivery to the Pelvic Floor Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Sebnem Alanya Tosun, Assistant Professor, Giresun University
Other Study IDs: Mode of Delivery
Record Dates: First submitted 2020-06-18; First posted 2020-07-16 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Incontinence; Pelvic Organ Prolapse
Keywords: pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Study group 1: Primiparous women who gave birth with ceserean section
- Study group 2: Primiparous women who gave birth with vaginal route delivery without episiotomy
- Study group 3: Primiparous women who gave birth with vaginal route delivery with episiotomy
- Control group: Nulliparous women

SUMMARY:
The childbirth is one of the risk factors for pelvic organ prolapse. In order to prevent the pelvic organ prolapse, the physicians do not routinely advice any exercises after deliveries. The investigators wondered if the mode of deliveries such as ceserean section, vaginal route delivery with episiotomy or vaginal route delivery without episiotomy effect the pelvic floor function differently or not. In order to evaluate this, the investigators are planning to measure the muscle tonus in primiparous women.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women 5-10 years after birth

Exclusion Criteria:

* Multiparous women Women with connective tissue disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only primiparous women
Study Population: 18-40 years old primiparous women who gave birth 5-10 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle tonus | 25.05.2020- 25.08.2020
  Pelvic floor muscle tonus is going to measure by vaginal perineometry.

SECONDARY OUTCOMES:
Female sexual function | 25.05.2020- 25.08.2020
  Female sexual function is going to evaluate by validated FSFI questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sebnem Alanya Tosun, Giresun, Turkey (Türkiye)